CLINICAL TRIAL: NCT03577860
Title: Evaluation of Variation of Ventilation and Pulmonary Aeration Using Electrical Impedance Tomography in Patients With Interscalene Brachial Plexus Block for Shoulder Surgery
Brief Title: Ventilation and Pulmonary Aeration, Electrical Impedance Tomography, Interscalene Brachial Plexus Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Henrique Cunha Ferraro, Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 48739315.4.0000.5505
Record Dates: First submitted 2018-06-06; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Brachial Plexus Block; Pulmonary Ventilation
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine 4ml (Active Comparator): The interscalene brachial plexus block is performed with 4ml at level of C5-6 roots
  Interventions: Drug: Bupivacaine 4 mL
- Bupivacaine 15ml (Active Comparator): The interscalene brachial plexus block is performed with 15ml at level of C5-6
  Interventions: Drug: Bupivacaine 15 mL

INTERVENTIONS:
Drug: Bupivacaine 4 mL — The interscalene brachial plexus block is performed with 4ml of bupivacaine-epinephrine 0,5%- 1:200,000
  Arms: Bupivacaine 4ml
Drug: Bupivacaine 15 mL — The interscalene brachial plexus block is performed with 15ml of bupivacaine-epinephrine 0,5%- 1:200,000
  Arms: Bupivacaine 15ml

SUMMARY:
Patients with indication of shoulder surgery will be submitted to ultrasound-guided interscalene brachial plexus block with 4ml or 15ml of bupivacaine- epinephrine 0,5%- 1:200,000 at level of C5-6 roots and will be evaluated their ventilation and pulmonary aeration by electrical impedance tomography

ELIGIBILITY:
Inclusion Criteria:

* shoulder surgery
* indication of interscalene brachial plexus block
* American Society of Anesthesiology Physical Status Classification I or II

Exclusion criteria:

* refuse to participate
* previous lung or diaphragma surgeries

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-10-17 (Estimated); Study Completion 2018-12-17 (Estimated)

PRIMARY OUTCOMES:
Variation of pulmonary function | 4 hour
  Evaluation of variation of pulmonary aeration and ventilation after interscalene brachial plexus block with 4ml or 15 ml of bupivacaine- epinephrine 0,5%1:200,0000. The pulmonary function will be evaluated by electrical impedance tomography.

SECONDARY OUTCOMES:
Opioid consumption | 24 hours
  Opioid consumption (Tramal - mg) will be recorded during the first 24 hours.
Post-Operative pain | 24 hours
  The post operative pain will be evaluated using Visual Analog Score for pain during the first 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo HC Ferraro, PhD, Principal Investigator — Federal University of São Paulo
Locations (2):
- Brazil (2):
  - Federal University of Sao Paulo, São Paulo
  - Federal University of Sao Paulo - Hospital Sao Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sinha SK, Abrams JH, Weller RS. Ultrasound-guided interscalene needle placement produces successful anesthesia regardless of motor stimulation above or below 0.5 mA. Anesth Analg. 2007 Sep;105(3):848-52. doi: 10.1213/01.ane.0000271912.84440.01. PMID 17717249
- [Result] Riazi S, Carmichael N, Awad I, Holtby RM, McCartney CJ. Effect of local anaesthetic volume (20 vs 5 ml) on the efficacy and respiratory consequences of ultrasound-guided interscalene brachial plexus block. Br J Anaesth. 2008 Oct;101(4):549-56. doi: 10.1093/bja/aen229. Epub 2008 Aug 4. PMID 18682410
- [Result] Gautier P, Vandepitte C, Ramquet C, DeCoopman M, Xu D, Hadzic A. The minimum effective anesthetic volume of 0.75% ropivacaine in ultrasound-guided interscalene brachial plexus block. Anesth Analg. 2011 Oct;113(4):951-5. doi: 10.1213/ANE.0b013e31822b876f. Epub 2011 Aug 4. PMID 21821517
- [Result] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Result] Urmey WF, McDonald M. Hemidiaphragmatic paresis during interscalene brachial plexus block: effects on pulmonary function and chest wall mechanics. Anesth Analg. 1992 Mar;74(3):352-7. doi: 10.1213/00000539-199203000-00006. PMID 1539813
- [Result] Renes SH, van Geffen GJ, Rettig HC, Gielen MJ, Scheffer GJ. Minimum effective volume of local anesthetic for shoulder analgesia by ultrasound-guided block at root C7 with assessment of pulmonary function. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):529-34. doi: 10.1097/AAP.0b013e3181fa1190. PMID 20975468
- [Result] Urmey WF, Gloeggler PJ. Pulmonary function changes during interscalene brachial plexus block: effects of decreasing local anesthetic injection volume. Reg Anesth. 1993 Jul-Aug;18(4):244-9. PMID 8398959
- [Result] Gottardis M, Luger T, Florl C, Schon G, Penz T, Resch H, Benzer A. Spirometry, blood gas analysis and ultrasonography of the diaphragm after Winnie's interscalene brachial plexus block. Eur J Anaesthesiol. 1993 Sep;10(5):367-9. PMID 11767428
- [Result] Hortense A, Perez MV, Amaral JL, Oshiro AC, Rossetti HB. Interscalene brachial plexus block. Effects on pulmonary function. Rev Bras Anestesiol. 2010 Mar-Apr;60(2):130-7, 74-8. doi: 10.1016/s0034-7094(10)70017-9. English, Portuguese, Spanish. PMID 20485957
- [Result] Renes SH, Rettig HC, Gielen MJ, Wilder-Smith OH, van Geffen GJ. Ultrasound-guided low-dose interscalene brachial plexus block reduces the incidence of hemidiaphragmatic paresis. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):498-502. doi: 10.1097/AAP.0b013e3181b49256. PMID 19920426